CLINICAL TRIAL: NCT01004133
Title: The Healthy Elderly Longevity Cohort
Acronym: Wellderly
Status: Recruiting | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute
Other Study IDs: HSC 07-4789
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Age 80 or older; No chronic disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — A single blood specimen or saliva specimen is collected from each subject. If blood is collected, approximately thirty eight milliliters of blood will be dispensed as follows:
  3 x 8.5 mls DNA Tubes
  1 x 2.5 mls RNA tube
  1 x 10 mls EBV tube (EDTA) for immortalized cell lines
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects 80 years of age or older without chronic diseases.

SUMMARY:
With the completion of the human genome project, investigators can now explore new questions in human biology. Previously human genetics focused on highly penetrant, Mendelian traits; however, now rare and common variants can be discovered that affect "common" diseases that have multi-gene architecture with variable penetrance such as breast cancer, diabetes mellitus, and coronary artery disease. This change took place because investigators now have the tools to illuminate the whole genome at once to discover the genetic variants responsible for different disease phenotypes through statistical differences between populations. Besides disease phenotypes, health can be considered a human phenotype that can be studied. Health is not merely the absence of disease but may be viewed as a dynamic ongoing interplay between the environment and the genome to maintain homeostasis. Individuals often attempt to optimize environmental conditions according to ones genome to maximize their health. All individuals possess potentially beneficial and harmful variants depending on the environment. How this dynamic interplay occurs between the genome and environment requires understanding the boundary conditions of the genetic architecture of health and disease and then modeling the system to simulate the observed data.

The aging process also affects health. Aging involves a loss of the normal coping responses to internal and external environmental stressors or signals. Investigators now have the tools to uncover from the bottom up the mechanisms involved in maintaining the ability to overcome environmental conditions that can affect health.

Against this genomic breakthrough of whole genome association studies, the demographics in the United States are quickly changing. The older population (age > 65 years) in 2030 is projected to be twice as large as in 2000 representing nearly 20 percent of the total US population. The first baby boomers turn 65 in 2011 and will challenge all facets of health care in the coming decades. The demographic changes underscore the need to understand the mechanisms that promote health and disease in this cohort. Genomic discoveries will help individuals and may reduce medical costs and benefit society.

In summary, the objective of this study is to obtain blood and/or saliva samples in order to help model health and disease phenotypes through population genomics. The blood and/or saliva samples may allow for participants' entire genomes to be sequenced if such comprehensive analysis becomes feasible and economical.

ELIGIBILITY:
Inclusion Criteria:

1. Age 80 years or older
2. Eligible for blood draw and/or saliva collection
3. Be reliable, cooperative and willing to comply with all protocol-specified procedures
4. Able to understand and grant informed consent
5. Be healthy or have mild medical conditions that may be associated with the normal aging process, including:

   * Hypertension, well controlled (no more than 3 medications)
   * Osteoporosis, Osteopenia and/or osteoarthritis
   * Benign prostatic hypertrophy
   * Cataracts, Glaucoma, Macular Degeneration
   * Dyslipidemia
   * Hypothyroidism
   * Pre-diabetes/impaired fasting glucose (fasting blood glucose 100-126 mg/dL, if known)

Exclusion Criteria:

1. < 80 years old
2. Participants have been previously enrolled in The Scripps Genebank Healthy Elderly Cohort
3. Treatment with any investigational agents or devices within thirty days preceding enrollment in the study.
4. Self-reported history or current diagnosis of significant chronic conditions including:

   * Any Cancer (including polycythemia; excluding basal or squamous cell skin cancer).
   * Coronary Artery Disease/Myocardial Infarction
   * Stroke/TIA
   * Deep Vein Thrombosis/Pulmonary Embolus
   * Chronic Renal Disease/Hemodialysis
   * Significant Auto-immune/Inflammatory conditions such as (Rheumatoid Arthritis, Lupus, Crohn's, etc.
   * Alzheimer's/Parkinson's
   * Diabetes (Hemoglobin A1C > 6.5 % or fasting glucose >126 mg/dL or treated with oral diabetic medication or insulin if known)
   * Aortic or Cerebral Aneurysm
5. Currently taking any of the following medications on a regular basis:

   * Oral chemotherapeutic agents (ex.: tamoxifen, doxorubicin, mitoxantrone, bleomycin)
   * Anti-platelet agents, not including aspirin (ex.: clopidogrel/plavix, dipyridamole/aggrenox/persantine, ticlopidine/ticlid)
   * Cholinesterase inhibitor for Alzheimer's disease (i.e. donepezil/Aricept)
   * Insulin
6. Subject has a significant medical condition which, in the Investigator's opinion, may interfere with the patient's optimal participation in the study or would potentially confound interpretation of the individual's phenotype.

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: General outpatient and community population.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2007-08; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Biorepository Creation | ten years
  Create a biorepository from participants' blood and/or saliva donations we will ultimately be able to define genes for various diseases and understand health

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States

REFERENCES:
- See also: Wellderly Study Web Site — https://www.scripps.edu/science-and-medicine/translational-institute/translational-research/genomic-medicine/wellderly/index.html?tab-1-text-content=1